CLINICAL TRIAL: NCT01380626
Title: Effects of Exercise Training on Quadriceps Gene Expression in COPD-patients in Comparison to Alpha-1-Antitrypsin-deficiency-patients
Brief Title: Effects of Exercise Training in Chronic Obstructive Pulmonary Disease Versus Alpha-1-Antitrypsin-deficiency-patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Grifols Therapeutics LLC (Industry); Alpha-1 Foundation (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician (department of pneumology), Schön Klinik Berchtesgadener Land
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AAT2010
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Alpha-1-antitrypsin-deficiency
Keywords: alpha-1-antitrypsin-deficiency; COPD; exercise training; muscle biopsy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; alpha 1-Antitrypsin Deficiency | interventions — Exercise; Endurance Training; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise training (Experimental)
  Interventions: Procedure: exercise training

INTERVENTIONS:
Procedure: exercise training — strength and endurance training, 5 time per week.
  Other Names: endurance training; strength training

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD)-patients (caused by smoking-level) and Alpha-1-Antitrypsin-deficiency patients showed different developments during rehabilitation in regard to improvement of 6-minute-walking distance. The aim of this study is to investigate differences between training adaptations in COPD-patients and Alpha-1-deficiency patients. Both groups take part in a standardized multimodal 3-week-rehabilitation with strength and endurance training. In addition to conventional diagnostic procedures, muscle biopsies from the M. vastus lateralis will be conducted before and after rehabilitation program followed by biochemical, histochemical and immunohistochemical analysis of the probes.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Alpha-1-Antitrypsine-deficiency, phenotype: ZZ
* FEV1%pred. <50

Exclusion Criteria:

* acute exacerbation
* exacerbation in the last 4 weeks

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
aerobic and anaerobic enzymes | day 2 and 23
  changes in quantity of enzymes from baseline to day 23

SECONDARY OUTCOMES:
maximal exercise capacity in incremental cycling test | day 2 and 23
  Change in max. exercise capacity from baseline to day 23
6-minute-walking distance | day 3 and 24
  change in 6-minute-walking distance from baseline to day 24

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Dr. med., Study Chair — Klinikum Berchtesgadener Land, Schön Klinik
Locations (1):
- Klinikum Berchtesgadener Land, Berchtesgaden, Germany